CLINICAL TRIAL: NCT00006216
Title: Treatment of Malignant Pleural Mesothelioma With Gene Modified Cancer Cell Lines
Brief Title: Vaccine Therapy and Ganciclovir in Treating Patients With Mesothelioma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068049; LSUMC-3591; NCI-V00-1604
Record Dates: First submitted 2000-09-11; First posted 2004-04-26 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-07

CONDITIONS: Malignant Mesothelioma
Keywords: stage IA malignant mesothelioma; stage IB malignant mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Ganciclovir

INTERVENTIONS:
Biological: PA-1-STK ovarian carcinoma vaccine
Drug: ganciclovir

SUMMARY:
RATIONALE: Ganciclovir may ease some of the side effects of cancer treatment. Vaccines made from a person's modified malignant mesothelioma cells may make the cancer more sensitive to ganciclovir.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy plus ganciclovir in treating patients who have stage I, stage II, or stage III malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and side effects of intrapleurally administered PA-1-STK modified ovarian carcinoma vaccine and ganciclovir in patients with stage I, II, or III malignant mesothelioma. II. Determine the maximum tolerated dose and dose limiting toxicities of this vaccine in these patients. III. Determine the immunologic response to this treatment regimen in these patients. IV. Determine the intrapleural pharmakokinetics of ganciclovir in these patients.

OUTLINE: This is a dose escalation study of PA-1-STK modified ovarian carcinoma vaccine. Patients receive PA-1-STK modified ovarian carcinoma vaccine intrapleurally on day 1 followed by ganciclovir IV over 1 hour for 7 days beginning on day 1. Patients in the first 2 cohorts receive 1 course of treatment only. In all subsequent cohorts, treatment repeats every 3 weeks for a total of 3 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3 patients receive escalating doses of PA-1-STK modified ovarian carcinoma vaccine until the maximum tolerated dose is determined.

PROJECTED ACCRUAL: A total of 3-16 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage I, II, or III malignant mesothelioma Must have adequate pleural space in which to place chest tube or catheter

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Hematocrit greater than 30% WBC greater than 4,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal SGOT and alkaline phosphatase less than 1.5 times normal Renal: Creatinine less than 1.5 mg/dL Creatinine clearance greater than 50 mL/min Cardiovascular: No significant history of heart disease No frequent angina No myocardial infarction within the past 6 months No congestive heart failure requiring daily treatment Pulmonary: No evidence of moderate to severe pulmonary disease (i.e., FEV1 less than 40% predicted) Other: No prior malignancy except squamous or basal cell carcinoma of the skin No patients with childbearing potential

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since prior chemotherapy Endocrine therapy: No concurrent steroid treatment Radiotherapy: At least 6 weeks since prior radiotherapy Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-08

CONTACTS AND LOCATIONS:
Overall Officials: Paul O. Schwarzenberger, MD, Study Chair — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Louisiana State University School of Medicine, New Orleans, Louisiana, United States